CLINICAL TRIAL: NCT03865875
Title: Pilot Study of a Multimodal Prehabilitation Pancreatic Cancer Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Motaz Qadan, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-635
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Ductal Adenocarcinoma; Total Neoadjuvant Therapy; Prehabilitation; Exercise; Nutrition; Optimization; Surgery
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training; Food Assistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimodal Prehabilitation Program (Experimental): Pretreatment exercise program and nutrition program
  -The prehabilitation intervention will include the following components: (1) a standardized fitness program and (2) nutritional counseling and optimization. Patients are enrolled in the program within 8 weeks of being diagnosed and continued until operation
  Interventions: Behavioral: Exercise Program; Behavioral: Nutrition Program

INTERVENTIONS:
Behavioral: Exercise Program — Participants will start the exercise program within 2 weeks of enrollment and will continue until surgery. This program will consist of twice weekly individualized sessions with a trainer.
Behavioral: Nutrition Program — Each patient enrolled will undergo nutritional assessment at their initial post-enrollment visit to develop an individualized nutrition plan to be implemented up until when the patient undergoes surgery.

SUMMARY:
The purpose of this research is to explore the benefits of an exercise and nutrition program during total neoadjuvant therapy (TNT) in preparation for surgery for participants that have pancreatic ductal adenocarcinoma (PDAC)

DETAILED DESCRIPTION:
This research study involves an exercise and nutrition program that will consist of twice weekly exercise sessions and discussion with a nutritionist with possible nutrition supplementation.

The names of the study interventions involved in this study are:

* Exercise Intervention
* Nutrition Intervention

The research study procedures include: screening for eligibility, study evaluations, and follow up visits.

ELIGIBILITY:
Inclusion Criteria

* Adults age 18 years or older.
* Diagnosed within 8 weeks with upfront resectable, borderline resectable, or locally advanced unresectable PDAC as defined by the National Comprehensive Cancer Network (NCCN).
* Planning to undergo TNT at MGH.
* Planning to receive modified FOLFIRINOX for neoadjuvant chemotherapy.
* Planning to undergo surgical resection of PDAC at MGH.
* Verbal fluency in English.

Exclusion Criteria

* Metastatic disease.
* Previous treatment for pancreas adenocarcinoma and no prior therapy for any cancer within 5 years.
* Known history of cognitive or psychologic impairment.
* Known history of physical impairment such as immobility, use of walking aids, or required wheelchair use.
* Known history of the following orthopedic comorbidities: advanced osteoarthritis or rheumatoid arthritis, mobility-limiting amputations, orthopedic injuries, or widespread chronic pain (e.g. fibromyalgia).
* Known history of the following pulmonary comorbidities: severe chronic obstructive pulmonary disease (COPD) defined as FEV1 ≤ 50%, emphysema, interstitial lung disease, and/or use of supplemental oxygen.
* Known history of the following cardiovascular comorbidities: uncontrolled hypertension, severe congestive heart failure (NYHA Class IV), and/or myocardial infarction within the last 6 months.
* Inability to tolerate diet through routine oral routes and/or patients with strict nutritional restrictions, allergies, and/or dietary preferences.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-13 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants to complete prehabilitation program | 1 year
  At least 50% (95% confidence interval +/- 16%) of participants will complete 50% of the components of the prehabilitation program.

CONTACTS AND LOCATIONS:
Overall Officials: Motaz Qadan, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation
URL: http://www.dfhcc.harvard.edu/crs-resources/ODQ_Documents/02_CT.GOV_CTRP/Guidance_on_Data_Sharing.pdf